CLINICAL TRIAL: NCT07297771
Title: Investigation of Latissimus Dorsi Muscle Activation During Different Exercises
Brief Title: Latissimus Dorsi Activity During Different Exercises
Acronym: L-DORSI-EMG
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Irem Duzgun, Professor, Department of Physiotherapy and Rehabilitation, Hacettepe University
Other Study IDs: LDORSI-EMG
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Muscle Activation
Keywords: Latissimus Dorsi; Shoulder; Electromyography
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy adults: Single-visit laboratory cohort. Physically active adults perform exercises; surface EMG is recorded from the latissimus dorsi
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Participants will perform six standardized pulling tasks-inferior glide, low row, seated row, bent-over row, seated press-up, and body lifting-using a resistance band or body weight. Each exercise is done for 3 repetitions with ~5 s between reps and ~2 min between exercises. Resisted exercises follow a metronome-paced 3 s concentric / 3 s isometric / 3 s eccentric tempo; purely isometric tasks are held for 3 s. Load is individualized with the OMNI 0-10 scale and increased during up to 10 familiarization reps until perceived exertion reaches 6-8/10. Exercise order is randomized to minimize ordering effects.

SUMMARY:
This single-visit, laboratory study will quantify latissimus dorsi activation during standardized band/body-weight exercises commonly used in rehabilitation (e.g., standing bent-over row, inferior glide, seated press-up, body-lifting). Healthy, physically active adults (18-40 y; Tegner ≥5) will perform three repetitions per exercise with metronome-paced phases (≈3 s concentric, 3 s isometric, 3 s eccentric), 5-s rest between repetitions and 2-min between exercises; load will be individualized to reach OMNI RPE 6-8. Surface EMG (TeleMyo DTS; Noraxon) will be recorded from the latissimus dorsi (medial and lateral) and selected synergists (teres major, infraspinatus, posterior deltoid, triceps); electrode placement will follow SENIAM recommendations. Signals will be band-pass filtered (20-500 Hz), rectified, RMS-smoothed with a 100-ms window, and normalized to %MVIC using standardized MVC tests; exercise/MVC order will be randomized to limit bias. The primary outcome is mean normalized EMG amplitude per exercise; secondary outcomes include peak amplitude and categorical activation levels (low ≤20% MVIC, moderate 21-40%, high 41-60%, very high >60%). The study involves minimal risk (possible mild skin irritation under electrodes and transient post-exercise fatigue).

DETAILED DESCRIPTION:
The latissimus dorsi (LD) originates from the spinous processes of the lower six thoracic vertebrae and the thoracolumbar fascia/iliac crest, and-together with the teres major-attaches to the medial lip of the intertubercular groove of the humerus. Functionally, LD contributes to shoulder adduction, internal rotation, and extension, linking the upper limb to the trunk. Alongside the rotator cuff, prevention of superior translation of the humeral head may be provided by the glenohumeral adductors (pectoralis major and LD) acting as humeral head depressors via a medio-inferior vector created by their tendon orientation. From an osteokinematic perspective, LD may protect against subacromial pain by facilitating inferior glide of the humeral head on the glenoid.

Selecting an appropriate strengthening exercise is critical to restore muscle performance and functional arm elevation in patients with shoulder injury or dysfunction. The literature emphasizes exercises targeting activation of the rotator cuff and scapulothoracic muscles that contribute to functional elevation. Surface electromyography (sEMG) is commonly used to guide exercise selection and progression by quantifying a muscle's contribution across different exercises, thereby enabling evidence-based advancement in strengthening programs.

However, much of the existing LD literature centers on lateral pull-down variations, with limited data for rehabilitation-relevant tasks such as low row, inferior glide, bent-over row (with trunk flexion), seated press-up, and body-lifting. Focusing on a single exercise limits clinical decision-making for shoulder rehabilitation (exercise selection and progression). Therefore, to support a scientific, evidence-based progression for LD strengthening in rehabilitation, this study was planned to obtain comprehensive sEMG data across multiple exercises.

Aim: To examine LD EMG activation levels during different exercises and determine between-exercise differences.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* No range-of-motion restriction at the glenohumeral joint
* No shoulder, cervical, or lumbar region complaints/injury within the past 6 months
* No systemic or neurological disease
* Competent to consent and provides written informed consent
* Tegner Activity Scale ≥ 5

Exclusion Criteria:

* Body mass index (BMI) > 25 kg/m²

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy, physically active adults aged 18-40 years. Eligibility requires Tegner ≥5, full glenohumeral range of motion, no shoulder/cervical/lumbar complaints in the past 6 months, and no systemic or neurological disease.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-10-12 (Actual); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Electromyography | Baseline (Day 1)
  Surface EMG from the latissimus dorsi (medial and lateral sites) will be recorded with an 8-channel system (TeleMyo DTS; Noraxon). Skin will be shaved and cleaned with 70% isopropyl alcohol; bipolar Ag/AgCl electrodes will be placed per SENIAM with a 2 cm inter-electrode distance (MLD ~lateral to T9; LLD ~4 cm inferior to the scapular inferior angle, midway between the spine and lateral trunk). A synchronized video (Logitech C920) will mark movement onset/offset and will be deleted after analysis (no copies kept). Signals will be normalized to %MVIC using three 5-s MVIC trials (30-s rest between trials; ~2-min between muscles) performed in standardized positions with verbal encouragement. The outcome is the mean %MVIC during the steady phase of each exercise.

SECONDARY OUTCOMES:
Electromyography-Other muscles | Baseline (Day 1)
  Surface EMG will also be recorded from teres major, infraspinatus, posterior deltoid, and triceps using the same preparation, SENIAM-based placement, and processing/normalization procedures described above. The outcome is the mean normalized EMG amplitude (%MVIC) during the steady phase of each exercise (isometric: central 3-s window; resisted: concentric 3 sec -isometric 3 sec- eccentric 3 sec).
Activity Level | Baseline (Day 1)
  Baseline physical activity will be characterized using the Tegner Activity Scale (0-10) prior to testing; higher scores indicate greater habitual activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Altındag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared. De-identified aggregate results will be disseminated in publications. The dataset includes physiological signals; synchronized videos are deleted after analysis.